CLINICAL TRIAL: NCT01030328
Title: Atorvastatin Plus Fenofibric Acid in the Reduction of Intermediate
Brief Title: AFRICA: Atorvastatin Plus Fenofibric Acid (TriLipix) in the Reduction of Intermediate Coronary Atherosclerosis
Acronym: AFRICA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of patient population
Sponsor: Piedmont Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: PH09001
Record Dates: First submitted 2009-11-04; First posted 2009-12-11 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Coronary Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TriLipix + Atorvastatin (Active Comparator): Two tables of TriLipix + Atorvastatin taken once a day by mouth.
  Interventions: Drug: TriLipix
- 2 (Placebo Comparator): 2 sugar pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 2 sugar pills by mouth once a day.
  Arms: 2
Drug: TriLipix — 135 mg of TriLipix + 40 mg of Atorvastatin by mouth once a day
  Arms: TriLipix + Atorvastatin

SUMMARY:
This study will examine how an approved drug (TriLipix), when used in combination with a statin (a drug that lowers blood cholesterol levels), affects the makeup of plaque. Patients will be randomly assigned to receive either the study treatment (TriLipix plus Atorvastatin) or the comparison treatment (a placebo). Comparison of the effect on the makeup of plaque will be done by using coronary artery computed tomography angiography (CTA), which all participants will have at enrollment and at the end of the study (18 months after enrollment).

DETAILED DESCRIPTION:
This study will examine how an approved drug (TriLipix), when used in combination with a statin (a drug that lowers blood cholesterol levels), affects the makeup of plaque. Comparison of the effect on the makeup of plaque will be done by using coronary artery CTA, which all participants will have at enrollment and at the end of the study.

Those who meet the eligibility criteria and sign the informed consent will be enrolled on study. Patients will be instructed on nutritional guidelines and other lifestyle changes for heart-healthy living.

If a patient has had a coronary CTA within the past two (2) months, they will not undergo the procedure at enrollment. If the patient has not had a coronary CTA within the past two (2) months, they will undergo a coronary CTA with contrast. Patients will be randomly assigned to receive either the study treatment (135 mg of TriLipix plus 40 mg of Atorvastatin) or the comparison treatment (a placebo or two pills that contains no active treatment). They will have a 50% chance of receiving the study treatment and a 50% chance of receiving the comparison treatment. This is a double-blind study, which means the patient, the research staff, and the physician will not know which treatment the patient is receiving. However, in case of an emergency, this information is immediately available to the physician.

Follow-up visits will occur at 3, 6, 12, and 18 months. All patients will have a CTA at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85
2. CAC 30-400, within 12 months of screening visit, OR intermediate stenosis on coronary artery CTA or invasive angiography (40-69% visual estimation) without the presence of obstructive (≥70% visual estimation) Stenosis within 3 months of screening visit
3. LDL-C ≥ 100 mg/dL and LDL-C ≤190 mg/dL at screening or baseline visit
4. TG>150 mg/dL and TG/HDL>3.5 at screening or baseline visit
5. 10 Year Framingham risk score of ≤ 10%
6. Ability and willingness to provide consent and Authorization for use of PHI

Exclusion Criteria:

1. Previous coronary revascularization (PCI, CABG)
2. Current lipid lowering therapy (includes statins, fibrates, niacin, omega 3 agents, intestinal cholesterol absorption inhibitors, cholestatic cholesterol absorption agents and other anti-lipemic agents.)
3. Known genetic form of hypercholesterolemia (e.g. familial hypercholesterolemia, etc.)
4. Creatinine 1.5 mg/dL or greater at baseline visit
5. Fasting serum triglycerides 500 mg/dL or greater at screening or baseline visit
6. Inability to perform CTA:

   1. Arrhythmia precluding diagnostic CT examination
   2. Known moderate or severe allergy to iodine-based contrast agents (mild prior reactions that could be treated as an outpatient or that could be prevented by pre-medication in the past do not constitute exclusion)
7. Uncontrolled hypertension (SBP>180 mmHg or DBP>130 mmHg on stable treatment)
8. Decompensated heart failure (NYHA class IV) at the time of enrollment
9. Known Pregnancy
10. Inability or unwillingness to consent and Authorization for use of PHI
11. Presence of any co-morbidity that makes life expectancy less than 24 months
12. Inability or unwillingness to comply with follow up procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in calcified plaque volume/percent, non-calcified high-density plaque volume/percent, and low-density plaque volume/percent | 18, 24, 30, and 36 months after initiation

SECONDARY OUTCOMES:
The secondary endpoint of the study will be the change in PAV of the "Study Lesion" from baseline to follow-up. PAV will be expressed as a ratio of the plaque volume/total vessel volume. | 24, 30, and 36 months after initiation

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Miller, MD, Principal Investigator — Piedmont Heart Institute
Locations (1):
- Piedmont Hospital, Atlanta, Georgia, United States